CLINICAL TRIAL: NCT06401967
Title: Feasibility, Acceptability, and Preliminary Outcomes of a Smartphone-Based Program for Reduction in Alcohol Consumption
Brief Title: Study of a Smartphone-Based Alcohol Reduction Program
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in research priorities
Sponsor: Pivot Health Technologies Inc. (Industry)
Responsible Party: Principal Investigator, Jennifer Marler, MD, VP of Clinical and Medical Affairs, Pivot Health Technologies Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C-510
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Alcohol Use, Unspecified
Keywords: alcohol reduction; digital health; mobile apps; health promotion
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Pivot Clear (Experimental): A program for alcohol reduction
  Interventions: Behavioral: Pivot Clear; Device: BACtrack breathalyzer

INTERVENTIONS:
Behavioral: Pivot Clear — A mobile app and program for alcohol reduction.
Device: BACtrack breathalyzer — Personal breathalyzer device that measures blood alcohol content.

SUMMARY:
Prospective, open label, single center clinical study enrolling up to 100 adult participants to evaluate the feasibility, acceptability, and preliminary outcomes of the Pivot Clear smartphone-based alcohol reduction program.

DETAILED DESCRIPTION:
This is a prospective, open label, single center clinical study conducted with institutional review board (IRB) approval enrolling up to 100 adult participants who report at-risk alcohol consumption behavior and would like to reduce or eliminate alcohol consumption. The study will be performed remotely on an ambulatory basis. Participants will be asked to set up and use the Pivot Clear program. The program includes an app, personal breathalyzer, and short message service (SMS) text-based coaching with an alcohol reduction specialist. The study duration is 52 weeks. While participants will have access to the program for 52 weeks, it is expected that for most participants, most active participation in the program will be complete by 12 weeks. The primary reporting time point will be 12 weeks, with expected passive, longer-term follow-up outcomes collected at 26 weeks and 52 weeks. Participants will receive online questionnaires at intervals throughout the study (baseline, weekly for the first 12 weeks, at 26 weeks and at 52 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Score of ≥ 3 for women and ≥ 4 for men on the AUDIT-C at screening
* Would like to reduce or eliminate alcohol consumption
* Resident of the United States
* Able to read and comprehend English
* Owns and uses a smartphone compatible with the study app (iPhone 6 and above, operating system iOS (iPhone operating system) 15 and above, or Android 7.0 and above, operating system Android 7.0 and above)
* Has daily internet access on smartphone
* Comfortable downloading and using smartphone apps
* Interested in working with an alcohol reduction coach via SMS text
* Willing to sign the Informed Consent Form (ICF)

Exclusion Criteria:

* Currently using other support to reduce or quit alcohol, including apps, coaching, support groups, classes or quit programs
* Pregnant (self-reported)
* Self-reported past or present diagnosis of Alcohol Use Disorder (AUD)
* Self-reported past or present diagnosis of Substance Use Disorder
* Current use of the following medications: suboxone, methadone, or daily use of a benzodiazepine [including Alprazolam (e.g., Xanax), lorazepam (e.g., Ativan), clonazepam (e.g., Klonopin), diazepam (e.g., Valium), and temazepam (e.g., Restoril)]
* History of hospitalization or in-patient treatment due to alcohol use
* Using other alcohol reduction or abstinence apps, coaching, support groups, classes, or programs at study entry
* Failure to provide contact or collateral information, and/or failure to verify email address
* Participation in a previous study sponsored by Pivot Health Technologies, Inc. (formerly Carrot Inc.)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who complete all 12 weekly follow-up assessments | 12 weeks
  Calculated as the number of participants who complete 12/12 of the weekly follow-up assessments (specifically during the first 12 weeks of the study), divided by the total number of enrolled participants.

SECONDARY OUTCOMES:
Trial feasibility - enrollment | Baseline
  Trial feasibility is assessed with multiple measures of enrollment success; all are the percentage of potential participants that remain eligible after each pre-enrollment step.
  1. The percent of potential participants who complete the online screening that are eligible for participation.
  2. The percent of potential participants who complete the eligibility phone call that are eligible for participation.
  3. The percent of potential participants who remain eligible after the screening call who consent and complete study enrollment (study enrollment includes: electronically signing the informed consent form, completing the baseline questionnaire, and completing registration in the app).
Trial feasibility - questionnaire completion | 52 weeks
  Trial feasibility is assessed with measuring the percent of enrolled participants who complete at least 80% of all study questionnaires.
Average weekly alcohol consumption | 1-12, 26, and 52 weeks
  Reported as the mean number of standard drinks per week over the past 7-28 days, based on the timeline follow-back (TLFB) calendar method.
Proportion of participants with average drinks per day ≤ 2/day for men and ≤ 1/day for women | 1-12, 26, and 52 weeks
  Based on the average weekly alcohol consumption which is reported as the mean number of standard drinks per week over the past 7-28 days, based on the timeline follow-back (TLFB) calendar method.
  Calculated as the number of participants with average drinks per day ≤ 2/day for men and ≤ 1/day for women over the specified time period, divided by the total number of enrolled participants.
Proportion of participants who complied with the low-risk guideline for problematic drinking | 1-12, 26, and 52 weeks
  The low-risk guideline for problematic drinking is defined as having consumed no more than 7 drinks per week and no more than 3 drinks on any single day (for women), or 14 drinks per week and no more than 4 drinks on any single day (for men).
  Based on the average weekly alcohol consumption which is reported as the mean number of standard drinks per week over the past 7-28 days, based on the timeline follow-back (TLFB) calendar method.
  Calculated as the number of participants meeting the above low-risk guideline criteria over the specified time period, divided by the total number of enrolled participants.
Average daily alcohol consumption | 1-12, 26, and 52 weeks
  Reported as the mean number of standard drinks per day over the past 7-28 days, based on the timeline follow-back (TLFB) calendar method.
Average drinks per drinking day | 1-12, 26, and 52 weeks
  Reported as the mean number of standard drinks per drinking day (excluding days where no drinks were consumed) over the past 7-28 days, based on the timeline follow-back (TLFB) calendar method.
Proportion of participants with an AUDIT-C score below the threshold for unhealthy alcohol use in the U.S. | 12, 26, and 52 weeks
  AUDIT-C = Alcohol Use Disorders Identification Test-Consumption (the first three questions from the 10-item AUDIT, a tool developed by the World Health Organization to evaluate a person's use of alcohol).
  AUDIT-C scores range from 0 to 12 points, and are a sum of scores for each of its 3 questions. Lower scores indicate less alcohol use; higher scores indicate greater alcohol use. Unhealthy alcohol use in the U.S. is defined as a score greater than 4 for men, and a score greater than 3 for women.
  The number of individuals that have AUDIT-C scores below these thresholds will be divided by the total number of participants to obtain this outcome proportion.
Proportion of participants who reduced their AUDIT-C score category by by ≥ 1 risk level | 12, 26, and 52 weeks
  AUDIT-C = Alcohol Use Disorders Identification Test-Consumption.
  AUDIT-C scores range from 0 to 12 points, and are a sum of scores for each of its 3 questions. Lower scores indicate less alcohol use; higher scores indicate greater alcohol use. Unhealthy alcohol use in the U.S. is defined as a score greater than 4 for men, and a score greater than 3 for women.
  AUDIT-C scores can also be categorized into four risk levels: 0-4 indicates lower risk, 5-7 indicates increasing risk, 8-10 indicates higher risk, and 11 to 12 indicates possible dependence. An example of reducing by one risk level: a change from a score of 6, "increasing risk", at baseline to a score of 3, "lower risk", at follow-up.
  The number of individuals that reduce their AUDIT-C score category by at least one risk level will be divided by the total number of participants to obtain this outcome proportion.
Proportion of participants with an AUDIT score within the "lower risk" category | 12, 26, and 52 weeks
  AUDIT = Alcohol Use Disorders Identification Test (10-items, a tool developed by the World Health Organization to evaluate a person's use of alcohol).
  AUDIT scores range from 0 to 40 points. The score is a sum of scores for its 10 questions, each of which range from 0 to 4. Lower scores indicate less alcohol use; higher scores indicate greater alcohol use. Scores of 8 and greater are suggestive of an alcohol problem.
  AUDIT scores can also be categorized into four risk levels: 0-7 indicates lower risk, 8-15 indicates increasing risk, 16-19 indicates higher risk, and 20+ indicates possible dependence. An example of reducing by one risk level: a change from a score of 9, "increasing risk", at baseline to a score of 5, "lower risk", at follow-up.
  The number of individuals that have AUDIT scores of 7 or lower will be divided by the total number of participants to obtain this outcome proportion.
Proportion of participants who reduced their AUDIT score category by by ≥ 1 risk level | 12, 26, and 52 weeks
  AUDIT = Alcohol Use Disorders Identification Test (10-items, a tool developed by the World Health Organization to evaluate a person's use of alcohol).
  AUDIT scores range from 0 to 40 points. The score is a sum of scores for its 10 questions, each of which range from 0 to 4. Lower scores indicate less alcohol use; higher scores indicate greater alcohol use. Scores of 8 and greater are suggestive of an alcohol problem.
  AUDIT scores can also be categorized into four risk levels: 0-7 indicates lower risk, 8-15 indicates increasing risk, 16-19 indicates higher risk, and 20+ indicates possible dependence. An example of reducing by one risk level: a change from a score of 9, "increasing risk", at baseline to a score of 5, "lower risk", at follow-up.
  The number of individuals that reduce their AUDIT score category by at least one risk level will be divided by the total number of participants to obtain this outcome proportion.
Number of heavy drinking days | 1-12, 26, and 52 weeks
  Heavy drinking days are defined as days with ≥ 5 drinks for men and ≥ 4 drinks for women.
  Based on the timeline follow-back (TLFB) calendar method; 7-day follow-back for weeks 1-12 and 28-day follow-back for weeks 26 and 52.
  The number of heavy drinking days will be determined by counting the number of days of heavy drinking within each follow-back period.
Maximum number of drinks on any day over the timeline follow-back period | 1-12, 26, and 52 weeks
  Based on the timeline follow-back (TLFB) calendar method; 7-day follow-back for weeks 1-12 and 28-day follow-back for weeks 26 and 52.
  The maximum number of drinks will be determined over the 7-day follow-back periods for weeks 1-12, and the 28-day follow-back periods for weeks 26 and 52.
Proportion of days abstinent | 1-12, 26, and 52 weeks
  Based on the timeline follow-back (TLFB) calendar method; 7-day follow-back for weeks 1-12 and 28-day follow-back for weeks 26 and 52.
  Proportion of days abstinent will be calculated as number of days where 0 drinks were reported that day, out of the total number of days in that follow-back period (7 or 28).
Average duration of continuous abstinence | 12, 26, and 52 weeks
  Based on the timeline follow-back (TLFB) calendar method; 7-day follow-back for weeks 1-12 and 28-day follow-back for weeks 26 and 52.
  Calculated as the average number of consecutive days where 0 drinks were reported on the timeline follow-back.
Proportion of participants who reduced their World Health Organization (WHO) risk drinking level by ≥ 1 risk level | 12, 26, and 52 weeks
  The WHO risk drinking levels are defined as follows:
  low risk = 0 to 2.9 drinks/day (men) and 0 to 1.4 drinks/day (women) medium risk = 3.0 to 4.3 drinks/day (men) and 1.5 to 2.8 drinks/day (women) high risk = 4.4 to 7.1 drinks/day (men) and 2.9 to 4.3 drinks/day (women) very high risk = 7.2+ drinks/day (men) and 4.4+ drinks/day (women)
  Based on the average daily alcohol consumption which is reported as the mean number of standard drinks per day over the past 7-28 days, based on the timeline follow-back (TLFB) calendar method. Example of reducing one drinking level: a woman decreasing from an average of 3 drinks per day (high risk) to an average of 2 drinks per day (medium risk).
  The number of individuals that reduce their WHO risk drinking level by at least one level will be divided by the total number of participants to obtain this outcome proportion.
Adverse consequence related to alcohol | 12, 26, and 52 weeks
  Adverse consequence related to alcohol are assessed via the short inventory of problems revised (SIP-R), a15-item measure. The 15 items are rated on a 4-point scale (from 0-3); 0 = Never, 1 = Once or a few times, 2 = Once or twice a week, 3 = Daily or almost daily.
  Scores for the SIP-R range from 0 to 45, where a higher score indicates experience with greater adverse consequences related to alcohol.
Drinking motivations | 12, 26, and 52 weeks
  Drinking motivations are assessed via the Drinking Motivation Questionnaire Revised (DMQR, 20 items). The 20 items are rated on a 5-point Likert scale (from 1-5); 1 = Almost Never/Never, 2 = Some of the time, 3 = Half of the time, 4 = Most of the time, 5 = Almost Always/Always.
  This scale has 5 items each for reflecting the following four categories of motives: social, coping, enhancement, and external social pressures.
  The DMQR yields four scale scores (between 5 and 25) reflecting each of these motives for drinking alcohol, where a higher score indicates greater frequency of the reason motivating them to drink alcohol.
Desire to change drinking habits | Baseline
  Participants are asked: "Do you have any desire to change your drinking habits?"
  With the following options to answer:
  * No, I'm comfortable with my current habits
  * No, I know I could drink a little less but I'm not motivated to change right now
  * Yes, I'm interested in drinking a little less
  * Yes, I'm interested in drinking a lot less
  * Yes, I'm interested in stopping drinking for a short period of time
  * Yes, I'm interested in stopping drinking for a long period of time
Reasons for desired change in drinking habits | Baseline
  Participants are asked: "What are your reasons for wanting to change your drinking?" The following options are provided (participants select all that apply): physical health/disease prevention or disease management, physical wellness/fitness, spend less money, diet/reduce calorie intake, mental health, mindfulness goals, relationship improvement, work/career improvement, or other (please describe).
  Participants are then asked to rank the selected options starting at 1 = Most important (ending at the number of reasons that were selected).
Readiness to change | 4 and 12 weeks
  Participants are asked: "How ready are you to make changes to your drinking habits?" Answered on a range from 1-10; 1 = not at all ready, 10 = extremely ready. A higher score indicates greater readiness to change drinking habits.
Expected success to change drinking habits | 4 and 12 weeks
  Participants are asked: "If you were to change your drinking habits now, how successful would you be?" Answered on a range from 1-10; 1 = not at all successful, 10 = extremely successful. A higher score indicates greater expected success in changing drinking habits.
Expected difficulty maintaining reduction/abstinence | 4 and 12 weeks
  Participants are asked: "If you were to change your drinking habits now, how difficult do you think it would be to keep your new habits?" Answered on a range from 1-10; 1 = not difficult at all, 10 = extremely difficult. A higher score indicates greater expected difficulty to change drinking habits.
Satisfaction with current drinking behavior | 12, 26, and 52 weeks
  Participants are asked: "How satisfied are you with your current drinking behavior?" Answered on a range from 1-10; 1 = not at all satisfied, 10 = very satisfied. A higher score indicates greater satisfaction with current drinking behavior.
User feedback - set up and getting started with the program | 4 weeks
  Assessed with the following question: "How easy or difficult was it to set-up and get started in the Pivot program?" Participants answer on a 1-10 scale; 1 = very difficult, 10 = very easy. A higher score indicates an easier time setting up and getting started with the program.
User satisfaction - Net Promoter Score | 4, 12, and 26 weeks
  Specifically regarding likelihood to recommend to a friend or colleague, Net Promoter Score (NPS). Participants are asked: "How likely would you be to recommend the Pivot Clear program to a friend or colleague that had a desire to drink less?" Answered on a range from 1-10; 1 = not at all likely, 10 = very likely. A higher score indicates greater user satisfaction and promotion of the program.
User satisfaction - how use of the program has affected alcohol consumption | 5 weeks
  Participants are asked: "How has using the Pivot program affected your alcohol consumption?"
  Participants are provided with the following options to choose from:
  * Using the program has increased my alcohol consumption
  * Using the program has not affected my alcohol consumption
  * Using the program has decreased my alcohol consumption
User satisfaction - effectiveness of the program | 12 weeks
  Participants are asked: "Did you find the Pivot Clear program effective so far?".
  Participants are provided 4 choices to answer: very effective, somewhat effective, not really effective, not at all effective
User satisfaction - whether the program helped the participant maintain alcohol reduction | 12, 26, and 52 weeks
  Participants are presented with the following statement: "The program has helped me maintain a new drinking level where I drink less than when I started the study." Participants are asked to select True/False.
User satisfaction - program's ability to help someone reduce or quit alcohol | 10 weeks
  Participants are asked: "Which of the following best describes the Pivot Clear program's ability to help someone reduce or quit alcohol?"
  Participants are provided the following options to choose from:
  * The program is extremely helpful
  * The program is helpful
  * The program does not affect being able to reduce or quit alcohol
  * The program makes reducing or quitting alcohol more difficult
User satisfaction - perceived need for the program | 4 weeks
  Participants are asked: "Which of the following best describes your need for the Pivot Clear program".
  Participants are provided the following options to choose from:
  * I really need this program
  * I somewhat need this program
  * I don't need this program
  * I am not at all interested in this program
User satisfaction - effect of program on motivation to reduce/abstain | 3 weeks
  Participants are asked: "How has using the Pivot program affected your motivation to change your drinking habits?"
  Participants are provided with the following options to choose from:
  * Using the program has increased my motivation to change my drinking habits
  * Using the program has not affected my motivation to change my drinking habits
  * Using the program has decreased my motivation to change my drinking habits
User feedback - initial reactions to program design, specific program features including the breathalyzer, coaching, lessons, and drink tracking | 1 week
  Participants are asked: "What best describes your initial reaction to finding out a [breathalyzer; coach; drink tracker] was a part of this program?"
  Participants are provided the following to choose from:
  * I thought it was out of place in the program as I think it is [a legal/compliance/negative tool for; a substance abuse counselor for; only used by] those with a severe drinking problem
  * I don't think it is necessary or helpful
  * I was curious about it and didn't have strong feelings
  * Made sense to me as this was a program related to [alcohol, behavior change, alcohol consumption behavior]
  * I was very interested to use it
User feedback - program design, specific program features including the breathalyzer, coaching, lessons, and drink tracking | 2, 3, 5, and 12 weeks
  Participants are asked various questions regarding program features and design.
  Participants are asked: "Have you gained any insights from your [initial use of the breathalyzer; initial interactions with the drink tracker in the Pivot app; initial interactions with the coach; interactions with the lessons]? Check all that apply."
  Participants are provided the following options to choose:
  * Not applicable
  * Not really
  * It confirmed what I already thought
  * It was motivating
  * It was demotivating
  * It triggered me to drink more
  * It triggered me to drink less
User satisfaction - aspects of program participant enjoyed most/least | 12 weeks
  Participants are asked: "What aspect of the program do you enjoy the most so far?" and "What aspect of the program do you enjoy the least so far?".
  For both questions they are provided the following to choose from:
  * Coaching
  * Tracker
  * Lessons
  * Breathalyzer
  * Other app contents/features (please specify)
User feedback - possible future program features | 12 weeks
  Participants are asked about potential future program features (small interest groups, breathalyzer connected to the app, text-based community, coaching via phone calls).
  They are provided the following to choose from:
  * Very interested
  * Somewhat interested
  * Probably not interested
  * Definitely not interested
  * Comments (optional)
Use of other alcohol reduction or abstinence tools (apps, counseling, medications, etc.) | 11, 26, and 52 weeks
  Assessed via self-report. Participants are asked about other alcohol reduction or abstinence tools they have used throughout the last 6 months. Tools asked about include: apps (other than Pivot), counseling, medications, acupuncture, hypnotherapy, etc. Participants can report other tools not included in the list provided. Outcome reported as the number of participants who have used each other alcohol reduction or abstinence tools.
Engagement with the program - app openings | 26 weeks
  Collected via back-end app data collection. Engagement is specifically assessed with number of times the Pivot app was opened (number of app openings), number of days the app was opened, and the number of weeks the app was opened. All are assessed over the first 26 weeks of study enrollment.
Engagement with program - number of days with app openings | 26 weeks
  Collected via back-end app data collection. Engagement is specifically assessed with the number of days over which the app was opened by participants over the first 26 weeks of study enrollment.
Engagement with program - number of weeks with app openings | 26 weeks
  Collected via back-end app data collection. Engagement is specifically assessed with the number of weeks over which the app was opened by participants over the first 26 weeks of study enrollment.
Engagement with program - average duration of app sessions | 26 weeks
  Collected via back-end app data collection. Engagement is specifically assessed with the average duration of app sessions completed by participants over the first 26 weeks of study enrollment. Outcome unit of measure = duration in minutes.
Engagement with program - use of app features | 26 weeks
  Collected via back-end app data collection. Engagement is specifically assessed with the use of app features (Lessons, Drink Logging, Crush a Craving, Challenges/Triggers, Goal Setting) by participants over the first 26 weeks of study enrollment. Reported as the number of times each app feature was used.
Engagement with program - average number of messages | 26 weeks
  Collected via back-end app data collection. Engagement is specifically assessed with average number of messages sent by coach to participant per week and average number of messages sent by participant to coach per week, over the first 26 weeks of study enrollment.
Engagement with program - average number of weeks with coach engagement | 26 weeks
  Collected via back-end app data collection. Specifically, the average number of weeks with at least one message sent from participant to coach over the first 26 weeks of study enrollment.
Change in ratings of self-reported health indicators | 12 and 26 weeks
  The following health indicators are assessed: sleep quality, nutrition/diet quality, weight management, ability to manage stress, physical fitness, mental health (anxiety, depression, bipolar as applicable), and chronic diseases (cardiovascular disease, diabetes, high blood pressure, asthma, COPD, acid reflux as applicable).
  COPD = chronic obstructive pulmonary disease
  Participants are asked to rate each of the above health indicators on a scale of 1-5; 1 = poor, 5 = excellent.
  Ratings at each timepoint are compared to the baseline score to determine their change.
Average rating of positive change experienced in self-reported health indicators | 12 and 26 weeks
  The following health indicators are assessed: sleep quality, nutrition/diet quality, weight management, ability to manage stress, physical fitness, mental health (anxiety, depression, bipolar as applicable), and chronic diseases (cardiovascular disease, diabetes, high blood pressure, asthma, COPD, acid reflux as applicable).
  Participants are asked to rate each based on if they experienced any positive change in that area due to reduced drinking; scale 1-5; 1 = not at all, 5 = very much. Greater scores on the scale indicate greater positive change experienced in that area of health.
  The ratings for each health indicator are averaged across participants to generate the average rating.
Depressive symptoms | 12, 26, and 52 weeks
  Assessed via the Center of Epidemiological Studies Depression Scale (CES-D) screening questionnaire, 10 items. A score is calculated from a sum of the 10 items. Possible scores on the scale range from 0-30. Higher scores indicate greater severity of depressive symptoms, a worse outcome.
Anxiety | 12, 26, and 52 weeks
  Anxiety is assessed via Generalized Anxiety Disorder 7-item scale (GAD-7). The following is asked regarding the 7 items: "Over the last two weeks, how often have you been bothered by the following problems?". The 7 items are rated on a 4-point scale (from 0-3); 0 = Not at all, 1 = Several days, 2 = More than half the days, 3 = Nearly every day.
  Scores for the GAD-7 range from 0 to 21, where a higher score indicates greater severity of anxiety, a worse outcome. The following are score ranges and their associated anxiety severity: 0-4 minimal anxiety, 5-9 mild anxiety, 10-14 moderate anxiety, and 15-21 severe anxiety.
Resilience | 12, 26, and 52 weeks
  Resilience is assessed via The Brief Resilience Scale (6-item, self-report measure).
  The 6 items are rated on a 5-point scale (from 1-5); 1 = Strongly disagree, 2 = Disagree, 3 = Neutral, 4 = Agree, 5 = Strongly agree.
  Scores for the Brief Resilience Scale range are a result of adding the scores for the 6 items together and dividing that total by 6 (this is the average score for the items). Scores range from 1 to 5, where a higher score indicates greater resilience, a better outcome.
Well-being | 12, 26, and 52 weeks
  Well-being is assessed via the WHO-5 Well-being Index (5 items) score.
  The 5 items are rated on a 6-point scale (from 5-0); 5 = All of the time, 4 = Most of the time, 3 = More than half the time, 2 = Less than half the time, 1 = Some of the time, 0 = At no time.
  Scores for the WHO-5 Well-being Index result from adding the scores for the 5 items together. The score ranges from 0 to 25, where a higher score indicates greater well-being and quality of life, a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Marler, MD, Principal Investigator — Pivot Health Technologies Inc.
Locations (1):
- Pivot Health Technologies, Inc., San Carlos, California, United States